CLINICAL TRIAL: NCT01482611
Title: Phase I, First-in-human, Double-blind, Randomized, Placebo-controlled Trial to Examine the Safety, Tolerability and Plasma Pharmacokinetics of Increasing Single Oral Doses of JNJ-47910382 in Healthy Caucasian and Japanese Volunteers
Brief Title: A Study in Healthy Participants Investigating the Safety, Tolerability and Plasma Pharmacokinetics (PK) of Single Oral Doses of JNJ-47910382
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR018547; 47910382HPC1001 (Other: Janssen R&D Ireland); 2011-003196-11 (EudraCT Number)
Record Dates: First submitted 2011-10-24; First posted 2011-11-30 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C Virus; JNJ-47910382; 47910382HPC1001; HCV; Hepatitis C; Hep C; Healthy participants; Japanese; Caucasians
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel 1: Caucasian (Experimental): 10, 75 and 300 mg JNJ-47910382 or placebo
  Interventions: Drug: JNJ-47910382; Drug: Placebo
- Panel 2: Caucasian (Experimental): 30, 150, 600 mg JNJ-47910382 or placebo
  Interventions: Drug: JNJ-47910382; Drug: Placebo
- Panel 3: Japanese (Experimental): Session VIII and X: Doses of JNJ-47910382 or placebo to be determined
  Interventions: Drug: JNJ-47910382; Drug: Placebo
- Panel 4: Japanese (Experimental): Session IX: Dose of JNJ-47910382 or placebo to be determined
  Interventions: Drug: JNJ-47910382; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-47910382 — Type = exact number, unit = mg, number = 10, 75, 300, form = suspension, route = oral use.
  Arms: Panel 1: Caucasian
Drug: JNJ-47910382 — Type = exact number, unit = mg, number = 30, 150, 600, form = suspension, route = oral use.
  Arms: Panel 2: Caucasian
Drug: JNJ-47910382 — Type = exact number, unit = mg, number = To be determined, form = suspension, route = oral use.
  Arms: Panel 3: Japanese
Drug: JNJ-47910382 — Type = exact number, unit = mg, number = To be determined, form = suspension, route = oral use.
  Arms: Panel 4: Japanese
Drug: Placebo — Type = exact number, unit = mg, number = equivalent of 10, 75, 300, form = suspension, route = oral use.
  Arms: Panel 1: Caucasian
Drug: Placebo — Type = exact number, unit = mg, number = equivalent of 30, 150, 600, form = suspension, route = oral use
  Arms: Panel 2: Caucasian
Drug: Placebo — Type = exact number, unit = mg, number = equivalent dose to be determined, form = suspension, route = oral use.
  Arms: Panel 3: Japanese
Drug: Placebo — Type = exact number, unit = mg, number = equivalent dose to be determined, form = suspension, route = oral use
  Arms: Panel 4: Japanese

SUMMARY:
The purpose of this study is to investigate the safety, tolerability and plasma pharmacokinetics (PK) of JNJ-47910382 after increasing single oral doses (taken with food) from 10 mg up to 600 mg or up to the maximum tolerated dose or up to the dose that yields a JNJ-47910382 plasma level that approaches the predefined maximum mean exposure (whichever comes first) in healthy Caucasian and Japanese participants. The foreseen maximum dose is 600 mg. In addition, the effect of fasting (ie JNJ-47910382 is taken without food) on the plasma pharmacokinetics of JNJ-47910382 after one selected oral dose given to healthy Caucasian participants will be studied. JNJ-47910382 is a drug that is being developed to treat Hepatitis C infection and is an inhibitor of the reproduction machinery of the Hepatitis C virus (HCV). Pharmacokinetics (PK) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
This is a Phase I, single-center, first-in-human, double-blind (neither the participant nor the investigator/medical staff knows whether placebo or JNJ-47910382 is given at a certain moment), randomized (treatment with placebo or JNJ-47910382 is assigned by chance), placebo-controlled trial in 18 healthy Caucasian and 16 healthy Japanese participants to investigate the safety, tolerability and plasma pharmacokinetics of single oral doses of JNJ-47910382. This trial consists of 3 Parts: 1. a single dose escalation part in healthy male and female Caucasians, 2. a single dose study investigating the effect of fasting in healthy male and female Caucasians and 3. a single dose escalation part in healthy male Japanese participants. Part 1 holds 6 sessions, each testing another dose of JNJ-47910382. Part 2 holds 1 session testing one dose and Part 3 holds 3 sessions, each testing another dose of JNJ-47910382. The doses pre-defined for the Caucasian cohort in Part 1 are 10 mg, 30 mg, 75 mg, 150 mg, 300 mg, and 600 mg, given in Session I till and including Session VI, respectively. These doses may be adjusted based on results obtained from previous sessions, but will not exceed 600 mg, the predefined maximal tolerated dose or a dose that yields a JNJ-47910382 plasma levels that approaches the predefined maximum mean exposure. The foreseen maximum dose is 600 mg.The doses for the Japanese cohort, given in Session VIII till and including Session X, respectively, and the dose for the fasting-session (Session VII) will be defined during the conduct of the study, based on the safety, tolerability and PK profiles obtained in the previously completed sessions. The Caucasian cohort is divided over 2 panels (Panel 1 and 2) of 9 participants, and to each Panel, 3 different doses are assigned, respecting a washout period of at least 10 days. The Japanese cohort is divided over 2 panels (Panel 3 and 4) of 8 participants and to Panel 3, 2 different doses are assigned, respecting a washout period of at least 10 days, and to Panel 4 only 1 dose of JNJ-47910382 is assigned. Either Panel 1 or 2 will be selected for the fasting-study Session, depending on the dose that has been selected for this fasting-study. Both, JNJ-47910382 and the placebo are liquids and will be administered in the mouth of the participants via an oral dispenser. The decision to escalate to the next dose in Part 1 and 3 will be taken with caution. After each session, the safety and tolerability (till and including 96h post dose) and the PK (till and including 24h post dose) results will be evaluated by the sponsor and principle investigator - in a blinded fashion. Only in case the previous dose is shown to be generally safe and tolerable and the maximum tolerated dose and the maximal mean plasma JNJ-47910382 levels have not been reached and the PK profile is satisfactory, the next session can start, using a selected and agreed dose. Safety evaluations between sessions include adverse events, vital signs (blood pressure and heart rate), electrocardiogram (ECG) (evaluation of the activity of the heart at certain time points), heart telemetry (continuous evaluation of the activity of the heart, for 12 hours), physical examination and clinical laboratory tests. Throughout the trial, in each session, the plasma PK profiles of JNJ-47910382 will be determined up to 96 hours after dosing. Also the amount of JNJ-47910382 recovered in the urine will be determined over 72 hours after intake of study medication in Session IV and in the Japanese Session with the same dose (either Session VIII, IX or X). A blood sample dedicated for the analysis of specific genes involved in the PK (metabolism) and transport of JNJ-47910382 will be collected from each participant, preferentially on Day-2 of one of the sessions. Also safety and tolerability of JNJ-47910382 will be determined throughout the trial. In each session a triplicate ECG is taken, vital signs are recorded, urinalysis is performed and biochemical and blood parameters are assessed on Days 1, 2 and 4. On Day3, vital signs are recorded and a triplicate ECG taken. On Day-1, a triplicate ECG is taken. Heart telemetric recordings are performed on Day-1 and Day1 for 12 hours. Physical examination occurs on Day-1 and Day5.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subjects between 18 and 45 years of age, inclusive.
* Japanese subjects between 20 and 45 years of age, inclusive.
* MALE Japanese subjects who has resided outside of Japan for no more than 5 years and whose parents and maternal and paternal grandparents are Japanese
* A body weight above 50 kg at screening
* Non-smoking for at least 3 months prior to screening

Exclusion Criteria:

* Female Caucasian, except if postmenopausal for at least 2 years or be surgically sterile.
* Hepatitis A, B or C infection
* Human Immunodeficiency Virus Type 1 (HIV-1) or Human Immunodeficiency Virus Type 2 (HIV-2) infection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events as a measure of safety and tolerability of JNJ-47910382 for each dose tested. | As of Day1 till and including 30-35 days after last drug intake
  Adverse Events (AEs) with onset during the treatment phase and AEs that have worsened since baseline will be analysed.
PK parameters after increasing single oral doses of JNJ-47910382, from 10 mg up to the maximum tolerated dose or up to 600 mg or up to the dose that yields a plasma level that approaches the predefined maximum mean exposure of JNJ-47910382. | Measured on Day1 till and including Day5 (i.e. predose, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 36h, 48h, 72h and 96h post dose) in each session.
  PK characteristics of JNJ-47910382 are determined based on plasma levels at one time point (Day3, 4 and 5), at 2 time points (Day2) and at 11 time points (Day1). Standard PK parameters such as Cmax (maximal concentration), Tmax (time point at moment maximal concentration is reached), AUClast (Area Under the Curve from time point of drug administration up to the last time point with a measurable concentration post dosing) etc. will be determined.
Change from baseline values for clinical laboratory parameters for each dose group. | On Day1, 2 and 4 during treatment, on Day of drop-out (i.e. from day of dosing in first session till 96h postdosing in last session) and on both Follow up visits (i.e. 10-14 days after last drug intake and 30-35 days after last drug intake).
Change from baseline values for ECG for each dose group. | On Day-1, 1, 2, 3 and 4 during treatment and on Day of drop-out (i.e. from day of dosing in first session till 96h postdosing in last session)..
Change from baseline values for vital signs for each dose group. | On Day1, 2, 3 and 4 during treatment and on Day of drop-out (i.e. from day of dosing in first session till 96h postdosing in last session) and on both Follow up visits (i.e. 10-14 days after last drug intake and 30-35 days after last drug intake).
Change from baseline values for physical examination for each dose group. | On Day-1, 4, Day of drop-out (i.e. from day of dosing in first session till 96h postdosing in last session) and on both Follow up visits (i.e. 10-14 days after last drug intake and 30-35 days after last drug intake).
Change from baseline values for cardia telemetry for each dose group. | Day1 (12 hours post-dose)
Percentage of participants with adverse events as a measure of safety and tolerability of JNJ-47910382 for each dose tested. | As of Day1 till and including 30-35 days after drop out (and Day of drop out can be from day of dosing in first session till 96h postdosing in last session)..
  AEs with onset during the treatment phase and AEs that have worsened since baseline will be analysed.

SECONDARY OUTCOMES:
Sequencing of genes that may affect safety, tolerability or PK of JNJ-47910382. | Per participant, once during the conduct of the study, preferentially on Day-2 of one of the sessions.
  Drug transporter genes OATP (organic anion transporting polypeptide) 1B1, OATP2B1, OATP1B3, ATP-binding cassette sub-family member ABCG2, ABCB1, multidrug resistance-associated protein MRP2 and bile salt export pump BSEP.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Neuss, Germany